CLINICAL TRIAL: NCT02760199
Title: 89Zr-AMG211 PET Imaging in Patients With Relapsed/Refractory Gastrointestinal Adenocarcinoma Before and During Treatment With AMG 211
Brief Title: 89Zr-AMG211 PET Imaging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150930
Record Dates: First submitted 2016-03-15; First posted 2016-05-03 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Advanced Gastrointestinal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 89Zr-AMG211 and 89Zr-AMG211 PET (Experimental)
  Interventions: Drug: 89Zr-AMG211; Device: 89-ZrAMG211 PET

INTERVENTIONS:
Drug: 89Zr-AMG211 — Injection of 89Zr-AMG211 for imaging.
Device: 89-ZrAMG211 PET — 89Zr-AMG211 PET scan(s).

SUMMARY:
AMG 211 is a bispecific single-chain antibody construct of the bispecific T-cell engager (BiTE®) class that targets human carcinoembryonic antigen (CEA, CD66e) on (tumor) cells and cluster of differentiation 3 (CD3) positive T-cells. AMG 211 is a potentially new targeted drug in the treatment of relapsed/refractory gastrointestinal adenocarcinoma, since those are CEA expressing tumors. A well-known challenge in current drug development using targeted therapies is the high level of heterogeneity of target expression that is present in specific tumor types. Radio-labeling of AMG 211 with the positron emission tomography (PET) radionuclide Zirconium-89 (89Zr) enables non-invasive imaging and quantification of AMG 211 distribution in cancer patients. By performing a 89Zr-AMG211 PET scan prior to treatment with AMG 211, the uptake of the tracer in the primary and metastatic tumor lesions and normal organ distribution can be evaluated. By performing a 89Zr-AMG211 PET scan during AMG 211 continuous intravenous (cIV) treatment the investigators will be able to evaluate the impact of prolonged steady state exposure of AMG 211 on tumor and tissue uptake. The 89Zr-AMG211 PET imaging study may help to identify patients more likely to benefit from AMG 211 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject will or is also participating in the ongoing phase 1 study in which AMG 211 is administered via cIV. 89Zr-AMG211 PET imaging will be performed before and/or during treatment with AMG 211 cIV
* Informed consent provided
* Male or Female ≥ 18 years of age at the time of informed consent
* Advanced relapsed/refractory gastrointestinal adenocarcinoma
* At least 1 measurable tumor lesion

  o In case the investigators do not find any uptake in metastatic liver lesions in the first set of patients on the 89Zr-AMG211 PET scan, than subsequent patients need to have at least 1 measurable tumor lesion outside the liver
* Archival tumor tissue available or is willing to undergo biopsy of a tumor lesion before the start of treatment
* Adequate hematological, renal, and liver function
* Body weight ≥ 45 kg
* Other inclusion criteria may apply

Exclusion Criteria:

* Malignancy other than GI adenocarcinoma requiring current therapy
* Evidence of uncontrolled systemic disease (other than GI adenocarcinoma), active infection, Hepatitis B and/or C, HIV, history of cardiac disease, history of significant central nervous system (CNS) disease, history of chronic autoimmune disease (with the exception of stable type 1 diabetes)
* Major surgery within 28 days of study day 1
* Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment in another investigational device or drug study. Other investigational procedures while participating in this study are excluded.

  o Exception to this criterion is the participation in the currently ongoing phase 1 study with AMG 211 cIV and all procedures related to this study.
* Treatment with any chemotherapy, radiotherapy, immunotherapy, biologic, or hormonal therapy for cancer within 14 days prior to study entry or not recovered from treatment
* Unresolved toxicities from prior anti-tumor therapy
* Males or Females of reproductive potential and unwilling to practice an acceptable method of effective birth control while on study through 30 days after receiving the last dose of study drug.
* Females who are pregnant, planning to become pregnant, lactating/breastfeeding or who plan to breastfeed while on study through 30 days after receiving the last dose of study drug
* Other exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
The quantitative uptake op 89Zr-AMG211 in tumor tissue, organs and blood circulation expressed in SUV (Standardized Uptake Value) | 1 year

SECONDARY OUTCOMES:
Response to AMG 211 therapy according to the immune related response criteria (irRC) will be correlated to 89Zr-AMG211 tumor uptake data (measured in SUV). | 1 year
Number of patients with adverse events after 89Zr-AMG211 injection as a measure of safety and tolerability. Incidence, nature and severity of adverse events (according to CTCAE version 4.03) will be measured. | 1 year

OTHER OUTCOMES:
Explore the target tissue saturation by AMG 211, defined as changes in tissue uptake of radioactivity concentration, and correlate it with pharmacokinetics. | 1 year
Evaluate 89Zr-AMG211 as a complementary tool for improved patient selection for targeted therapy with AMG 211. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: E. G.E. de Vries, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - VUmc, Amsterdam
  - University Medical Center Groningen, Groningen